CLINICAL TRIAL: NCT02585466
Title: Precise Quantification of Surrogate Nociception Measures "Bispectral Index (sBIS)-Electromyography (sEMG) Variabilities" and "Response Entropy-State Entropy (RE-SE) Difference". A Practice Alignment Study.
Brief Title: BIS and Entropy Nociception Monitoring
Acronym: BIS4
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Ashraf Dahaba, MD, Doz. Dr., Medical University of Graz
Other Study IDs: MUGraz4
Record Dates: First submitted 2015-10-16; First posted 2015-10-23 (Estimated); Last update posted 2015-10-26 (Estimated); Status verified 2015-10

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- BIS25: BIS 25 levels were subsequently maintained via propofol TCI 0.2 microg mL-1 TCI adjustments. Stable BIS values that showed no further decline and remained within BIS ±5 ofBIS 25 of the previous BIS value were considered an indicator of pseudo-steady state plasma effect-site equilibration
- BIS50: BIS 50 levels were subsequently maintained via propofol TCI 0.2 microg mL-1 TCI adjustments. Stable BIS values that showed no further decline and remained within BIS ±5 of either BIS 50 levels of the previous BIS value were considered an indicator of pseudo-steady state plasma effect-site equilibration

SUMMARY:
Reports have been appearing in literature over the past years of various nociception-antinociception monitors, introduced and promoted from major manufactures. Recently a new term Practice misalignment" has been recently coined indicating research study groups that are distant from daily anesthesia practice, with some scientific relevance but very little clinical relevance simulating "purely hypothetical" conditions that are not related to "everyday" anesthesia practice.

DETAILED DESCRIPTION:
Background: Reports have been appearing in literature over the past years of various nociception-antinociception monitors, introduced and promoted from major manufactures. Recently a new term Practice misalignment" has been recently coined indicating research study groups that are distant from daily anesthesia practice, with some scientific relevance but very little clinical relevance simulating "purely hypothetical" conditions that are not related to "everyday" anesthesia practice. These proposed new nociception-antinociception parameters are assumed to be "immune" from confounding factors commonly encountered such as neuromuscular block, remifentanil, or cardiovascular haemodynamically active drugs.

Methods: Investigators sought to quantify the basic components of these new nociception-antinociception parameters in response to various noxious stimuli, and then test them against the most confounding factors namely neuromuscular blocking agents (NMBAs) for sEMG, remifentanil analgesia and haemodynamic changes, while at the same time analysing the EEG and blood levels. Investigators examined two nociception -antinociception parameters basic components sBIS/sEMG and Response Entropy-State Entropy difference from the two main manufacturers GE and Medtronic.

Fifty patients, aged 18-65 years, undergoing general surgery on the lower limb were randomly allocated to the BIS 25 or BIS 50 groups. Exclusion criteria included alcohol or drug abuse, chronic treatment with antihypertensive or cardiovascular medications including β-blockers, and medications acting on the central nervous system such as benzodiazepines, antiepileptic and neuroleptic medications, After capnographic verification of proper lungs ventilation with 40% oxygen in air, either BIS 50 levels or BIS 25 were subsequently maintained via propofol TCI 0.2 microg mL-1 TCI adjustments. Stable BIS values that showed no further decline and remained within BIS ±5 of either BIS 50 levels or BIS 25 of the previous BIS value were considered an indicator of pseudo-steady state plasma effect-site equilibration. Two silver/silver chloride surface stimulating electrodes were placed 4 cm apart on the ulnar nerve at the wrist and connected to Innervator NS272 (Fisher & Paykel, Auckland, New Zealand) peripheral nerve stimulator. The ulnar nerve was stimulated in an ascending sequence of single twitch electric stimulations starting from 10 mA, up till 80 mA for a period of 10 s with a 3 min period between stimulations. BIS and Entropy data were recorded. After which patients were re-stimulated under remifentanil and again re-stimulated under NMBAs.

ELIGIBILITY:
Inclusion Criteria:

1. age 18-65 years

Exclusion Criteria:

1. Alcohol or drug abuse,
2. chronic treatment with antihypertensive or cardiovascular medications
3. medications acting on the central nervous system such as benzodiazepines, antiepileptic neuroleptics

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Fifty patients, aged 18-65 years, undergoing general surgery on the lower limb were randomly allocated to the BIS 25 or BIS 50 groups
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2008-04; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
BIS (Bispectral Index) variability | 3 minutes following a 10 seconds stimulation
  Bispectral Index (BIS) difference between the highest and lowest values

SECONDARY OUTCOMES:
EMG variability | 3 minutes following a 10 seconds stimulation
  Electromypgraphy (EMG) difference between the highest and lowest values
Response Entropy - State Entropy difference (RE-SE) | 3 minutes following a 10 seconds stimulation
  Difference between Respnse Entropy value (RE, derived from electroencephalography and electromyography) minus State Entropy (SE, derived from electroencephalography only)

REFERENCES:
- [Background] Viertio-Oja H, Maja V, Sarkela M, Talja P, Tenkanen N, Tolvanen-Laakso H, Paloheimo M, Vakkuri A, Yli-Hankala A, Merilainen P. Description of the Entropy algorithm as applied in the Datex-Ohmeda S/5 Entropy Module. Acta Anaesthesiol Scand. 2004 Feb;48(2):154-61. doi: 10.1111/j.0001-5172.2004.00322.x. No abstract available. PMID 14995936
- [Background] Sigl JC, Chamoun NG. An introduction to bispectral analysis for the electroencephalogram. J Clin Monit. 1994 Nov;10(6):392-404. doi: 10.1007/BF01618421. PMID 7836975
- [Background] Dahaba AA. Different conditions that could result in the bispectral index indicating an incorrect hypnotic state. Anesth Analg. 2005 Sep;101(3):765-773. doi: 10.1213/01.ane.0000167269.62966.af. PMID 16115989